CLINICAL TRIAL: NCT03959345
Title: Multicenter, Randomised, Open-label Phase III-IV Study to Evaluate the Efficacy of Cloxacillin and Fosfomycin Combination Versus Cloxacillin Monotherapy in Patients With Methicillin-susceptible Staphylococcus Aureus Bacteraemia: SAFO Trial
Brief Title: Efficacy of Cloxacillin and Fosfomycin Combination Versus Cloxacillin Monotherapy in Patients With MSSA Bacteremia
Acronym: SAFO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Data safety and monitoring board(DSMB) have been performed when half of sample size (SS)have been reached. Recruitment was slower than expected so SS was recalculated. After analysis of data, DSMB recommended to stop study.
Sponsor: Miquel Pujol (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Miquel Pujol, Principal Investigator, Medical Doctor, Institut d'Investigació Biomèdica de Bellvitge
Organization: Institut d'Investigació Biomèdica de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001207-37
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Methicillin Susceptible Staphylococcus Aureus Septicemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy group (Experimental): intravenous cloxacillin 2g/4h and fosfomycin 3 g/6h for the duration of 7 days treatment
  Interventions: Drug: Combination therapy group
- Standard therapy group (Active Comparator): intravenous cloxacillin 2g/4h for the duration of 7 days IV treatment
  Interventions: Drug: Standard therapy group

INTERVENTIONS:
Drug: Combination therapy group — Adult patients with MSSA bacteraemia will be randomized to Combination therapy group: patients will receive intravenous cloxacillin 2g/4h and fosfomycin 3 g/6h for the duration of 7 days treatment. After the first week, antibiotic treatment and duration will be decided by responsible clinician following clinical practice.
  Arms: Combination therapy group
Drug: Standard therapy group — Adult patients with MSSA bacteraemia will be randomized to Standard therapy group: patients will receive intravenous cloxacillin 2g/4h for the duration of 7 days IV treatment. After the first week, antibiotic treatment and duration will be decided by responsible clinician following clinical practice.
  Arms: Standard therapy group

SUMMARY:
Background: Despite management improvement in lasts years, S.aureus bacteremia leads to high morbidity and mortality. For over 50 years, methicillin-susceptible S.aureus (MSSA) bacteremia standard treatment was cloxacillin. Previous studies using different therapies and combination treatment fall to improve survival in these patients.

Aim: to demonstrate the efficacy of the cloxacillin and fosfomycin combination administered during the first week of treatment, compared with cloxacillin monotherapy in patients with MSSA bacteremia in treatment success. Methods: A multicentre, superiority, open-label, randomized, phase IV-III, two-armed parallel (1:1) groups clinical trial. Adult patients with MSSA bacteremia will be randomized to Combination therapy group: patients will receive intravenous cloxacillin 2g/4h and fosfomycin 3 g/6h for the duration of 7 days treatment, or Standard therapy group: patients will receive intravenous cloxacillin 2g/4h for the duration of 7 days IV treatment. After the first week, antibiotic treatment and duration will be decided by responsible clinician following clinical practice.

The primary endpoint is the treatment success measured at day 7 of treatment; a composite endpoint defined by all of the following criteria met after randomization: patient alive at day 7 AND stable or improved quick SOFA score (compared with baseline) at day 7 AND fever resolved at day 7 AND negative blood cultures for S. aureus at day 7.

In case of achieving statistical differences in the primary endpoint, investigators will perform a hierarchical analysis of the treatment success at Test of Cure visit (TOC, 12 weeks after randomization), defined by the presence of all of the following: patient alive at TOC AND no evidence of microbiological treatment failure defined as isolation of S. aureus from blood culture or other sterile site from day 8 after randomization until TOC.

Investigators have assumed a 74% of treatment success in monotherapy group. Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 183 subjects are necessary in first group and 183 in the second to find a statistically significant difference of 12%. It has been anticipated a drop-out rate of 5%.

Discussion: Randomized studies assessing efficacy of different treatment in MSSA bacteremia are lacking. This study could help to improve knowledge about MSSA bacteremia and whether combined treatment with cloxacillin and fosfomycin could improve outcomes compared with standard treatment.

DETAILED DESCRIPTION:
SAFO trial is a multicentre, superiority, open-label, randomized, phase IV-III, two-armed parallel (1:1) groups clinical trial comparing combination treatment with fosfomycin and cloxacillin with standard therapy with cloxacillin in adult patients with MSSA bacteremia.

Patients will be randomized to:

* Standard treatment group: patients will receive intravenous cloxacillin 2g/4h for the duration of 7 days IV treatment. If creatinine clearance is <30 mL/min cloxacillin will be administrated at dose of 2g every 6 hours.
* Combination therapy group: patients will receive intravenous cloxacillin as explained above and fosfomycin 3 g/6h for the duration of 7 days treatment. In case of renal failure, fosfomycin will be administrated as follow:

Creatinine clearance (mL/min) Fosfomycin dosage >40 3 g every 6 hours 20-40 3 g every 12 hours 10-20 3g every 24 hours <10 3 g every 48 hours Haemodialysis 3 g after haemodialysis Continuous renal replacement therapy 3 g every 24h hours

The duration of overall antibiotic treatment and the duration of intravenous treatment will be determined according to clinical criteria depending on status (complicated or uncomplicated bacteremia, source of infection) by responsible clinician according with current guidelines. Patient with complicated bacteremia will receive at least 4-6 week of antibiotic treatment.

Primary endpoint

Treatment success at day 7 is a composite outcome defined by all of the following criteria met after randomization:

* Patient alive at day 7 AND
* Clinical improvement measured by stable or improved quick SOFA score (compared with baseline) at day 7 AND
* Fever resolved at day 7 AND
* Negative blood cultures for S. aureus at day 7.

In case of statistical differences observed between groups in the primary endpoint, investigators will perform a hierarchical testing analyzing the treatment success at Test of Cure (TOC visit, 12 weeks after randomization).

Treatment success at TOC visit is defined by presence of all of the following:

* Patient alive at TOC;
* No isolation of MSSA in blood culture or in another sterile site from day 8 until Test of Cure visit (TOC, 12 weeks after randomisation). In case of patients with prolonged course of antibiotic treatment (more than 10 weeks), TOC visit will be performed two weeks after the end of treatment (EOT).

Treatment failure is defined by the presence of one of the following condition: all-cause mortality at TOC, positive blood cultures at day 7 or later, withdraw of the study because of adverse events related to study treatment, requirement of an additional MSSA-active antibiotic until day 7, lacking of clinical improvement at day 7.

Secondary endpoint

Clinical secondary endpoints:

* To compare all-cause mortality at days 7, 14, EOT and 90 after randomization in cloxacillin treatment group versus cloxacillin and fosfomycin treatment group.
* To evaluate persistent bacteremia (at least one positive blood culture) at day 3 and persistent bacteremia at day 7 after randomization in the two arms of treatment.
* To determine the microbiological relapse as defined by at least one positive blood culture for MSSA at least 72 hours after a preceding negative culture in the two arms of treatment.
* To evaluate microbiological treatment failure as defined by positive sterile site culture for MSSA at least 14 days after randomisation in the two arms.
* To determine the number of patients with persistent and relapsing bacteremia in the two arms of treatment.
* To evaluate the number of patients with complicated bacteremia, defined by persistent bacteremia, endocarditis or metastatic emboli, prosthetic devices) in the two arms of treatment.
* To determine the length of stay in intensive care unit and in hospital in both arms of treatment.
* Duration of intravenous antibiotic treatment. Sub group analysis for patients at high risk (persistent bacteraemia, metastatic infection, unknown focus of bacteraemia, endocarditis, pneumonia).

Microbiological secondary endpoints:

* To determine emergency of fosfomycin-resistant strains during therapy in the arm of combination treatment.
* To evaluate operon agr functionality and its relationship with Minimum Inhibitory Concentration (MIC) changes to vancomycin (VAN) and daptomycin (DAP) and with biofilm production.
* To analyze VAN and DAP MIC as markers of complications during bacteraemia.
* To determine the "in vitro" cloxacillin plus fosfomycin combination synergy.
* To realize whole genome sequencing and its changes in patients with treatment failure.

Pharmacological secondary endpoints:

* To determine minimum and maximum concentration in steady state of fosfomycin and cloxacillin.
* To evaluate pharmacokinetic variability of these concentration.
* To study the association between PK parameters and efficacy.

Security secondary endpoints:

To evaluate the security of cloxacillin and fosfomycin combination compared with cloxacillin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, aged ≥ 18 years;
* MSSA bacteraemia: ≥ 1 positive blood culture(s) for MSSA in the first 72 h up to randomisation in patients with clinical suspicion of infection;
* Written informed consent of the participant or the legal representative.

Exclusion Criteria:

* Severe clinical status with expected death <48h.
* Severe hepatic cirrhosis (Child-Pugh C).
* Moderate-severe cardiac chronic failure (NYHA III-IV).
* Prosthetic endocarditis (need for concomitant antibiotic therapy active against S. aureus together with the study antibiotics for the first 7 days of the study).
* No pre-existing evidence of S. aureus fosfomycin non-susceptibility.
* Known hypersensitivity to cloxacillin or fosfomycin.
* Polymicrobial bacteraemia with more than one microorganism in blood cultures.
* A positive pregnancy test or pregnancy or lactation at the time of inclusion.
* Miastenia gravis.
* Participation in another clinical trial.
* Previous participation in the present clinical trial.
* Acute SARS-CoV2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Treatment success at day 7 | Day 7 after randomization.
  Composite endpoint defined by all of the following criteria met after randomization: patient alive at day 7 AND stable or improved quick SOFA score (compared with baseline) at day 7 AND fever resolved at day 7 AND negative blood cultures for S. aureus at day 7.
Treatment success at TOC | 12 weeks after randomization
  In case of achieving statistical differences in the primary endpoint, we will perform a hierarchical analysis of the treatment success at Test of Cure visit (TOC, 12 weeks after randomisation).
  Treatment success at TOC visit, defined by presence of all of the following:
  * Patient alive at TOC;
  * No isolation of MSSA in blood culture or in another sterile site from day 8 until TOC.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Pujol Rojo, MD, PhD, Principal Investigator — Hospital Universitari Bellvitge
Locations (17):
- Spain (17):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan Despí Moisés Broggi, Sant Joan Despí, Barcelona
  - University Hospital Cruces, Barakaldo
  - Bellvitge University Hospital, Barcelona
  - Hospital del Mar, Barcelona
  - University Hospital Clínic de Barcelona, Barcelona
  - University Hospital Santa Creu i Sant Pau, Barcelona
  - University Hospital Arnau de Vilanova, Lleida
  - University Hospital Lucus Agustí, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Sant Joan, Reus
  - Corporació Sanitària Parc Taulí, Sabadell
  - University Hospital Virgen Macarena, Seville
  - University Hospital Joan XXIII, Tarragona
  - University Hospital Mùtua de Terrassa, Terrassa
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. We would wish to make our results available both to the community of scientists interested in infectious diseases and the biology of Staphylococcus aureus to avoid unintentional duplication of research.
  The preliminary results will be presented at international and national infectious diseases conferences and will be published in peer-reviewed journals. The results will also be made available through press and social media communications. Any formal presentation or publication of data collected from this study will be considered as a joint publication by the participating investigators and will follow the recommendations of the ICMJE. Individual participant data that underlie the results, after deidentification will be available. Proposals should be directed to the corresponding author.
Supporting Information: Study Protocol
Time Frame: immediately following publication and ending 5 years following article publication
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.

REFERENCES:
- [Background] Bergin SP, Holland TL, Fowler VG Jr, Tong SYC. Bacteremia, Sepsis, and Infective Endocarditis Associated with Staphylococcus aureus. Curr Top Microbiol Immunol. 2017;409:263-296. doi: 10.1007/82_2015_5001. PMID 26659121
- [Background] van Hal SJ, Jensen SO, Vaska VL, Espedido BA, Paterson DL, Gosbell IB. Predictors of mortality in Staphylococcus aureus Bacteremia. Clin Microbiol Rev. 2012 Apr;25(2):362-86. doi: 10.1128/CMR.05022-11. PMID 22491776
- [Background] Gasch O, Camoez M, Dominguez MA, Padilla B, Pintado V, Almirante B, Molina J, Lopez-Medrano F, Ruiz E, Martinez JA, Bereciartua E, Rodriguez-Lopez F, Fernandez-Mazarrasa C, Goenaga MA, Benito N, Rodriguez-Bano J, Espejo E, Pujol M; REIPI/GEIH Study Groups. Predictive factors for mortality in patients with methicillin-resistant Staphylococcus aureus bloodstream infection: impact on outcome of host, microorganism and therapy. Clin Microbiol Infect. 2013 Nov;19(11):1049-57. doi: 10.1111/1469-0691.12108. Epub 2013 Jan 17. PMID 23331461
- [Background] Minejima E, Mai N, Bui N, Mert M, Mack WJ, She RC, Nieberg P, Spellberg B, Wong-Beringer A. Defining the Breakpoint Duration of Staphylococcus aureus Bacteremia Predictive of Poor Outcomes. Clin Infect Dis. 2020 Feb 3;70(4):566-573. doi: 10.1093/cid/ciz257. PMID 30949675
- [Background] Gudiol F, Aguado JM, Almirante B, Bouza E, Cercenado E, Dominguez MA, Gasch O, Lora-Tamayo J, Miro JM, Palomar M, Pascual A, Pericas JM, Pujol M, Rodriguez-Bano J, Shaw E, Soriano A, Valles J. Diagnosis and treatment of bacteremia and endocarditis due to Staphylococcus aureus. A clinical guideline from the Spanish Society of Clinical Microbiology and Infectious Diseases (SEIMC). Enferm Infecc Microbiol Clin. 2015 Nov;33(9):625.e1-625.e23. doi: 10.1016/j.eimc.2015.03.015. Epub 2015 May 1. PMID 25937457
- [Background] Thwaites GE, Scarborough M, Szubert A, Nsutebu E, Tilley R, Greig J, Wyllie SA, Wilson P, Auckland C, Cairns J, Ward D, Lal P, Guleri A, Jenkins N, Sutton J, Wiselka M, Armando GR, Graham C, Chadwick PR, Barlow G, Gordon NC, Young B, Meisner S, McWhinney P, Price DA, Harvey D, Nayar D, Jeyaratnam D, Planche T, Minton J, Hudson F, Hopkins S, Williams J, Torok ME, Llewelyn MJ, Edgeworth JD, Walker AS; United Kingdom Clinical Infection Research Group (UKCIRG). Adjunctive rifampicin for Staphylococcus aureus bacteraemia (ARREST): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Feb 17;391(10121):668-678. doi: 10.1016/S0140-6736(17)32456-X. Epub 2017 Dec 14. PMID 29249276
- [Background] Grillo S, Cuervo G, Carratala J, Grau I, Pallares N, Tebe C, Guillem Tio L, Murillo O, Ardanuy C, Dominguez MA, Shaw E, Gudiol C, Pujol M. Impact of beta-Lactam and Daptomycin Combination Therapy on Clinical Outcomes in Methicillin-susceptible Staphylococcus aureus Bacteremia: A Propensity Score-matched Analysis. Clin Infect Dis. 2019 Oct 15;69(9):1480-1488. doi: 10.1093/cid/ciz018. PMID 30615122
- [Background] Grabein B, Graninger W, Rodriguez Bano J, Dinh A, Liesenfeld DB. Intravenous fosfomycin-back to the future. Systematic review and meta-analysis of the clinical literature. Clin Microbiol Infect. 2017 Jun;23(6):363-372. doi: 10.1016/j.cmi.2016.12.005. Epub 2016 Dec 9. PMID 27956267
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Derived] Grillo S, Pujol M, Miro JM, Lopez-Contreras J, Euba G, Gasch O, Boix-Palop L, Garcia-Pais MJ, Perez-Rodriguez MT, Gomez-Zorrilla S, Oriol I, Lopez-Cortes LE, Pedro-Botet ML, San-Juan R, Aguado JM, Gioia F, Iftimie S, Morata L, Jover-Saenz A, Garcia-Pardo G, Loeches B, Izquierdo-Cardenas A, Goikoetxea AJ, Gomila-Grange A, Dietl B, Berbel D, Videla S, Hereu P, Padulles A, Pallares N, Tebe C, Cuervo G, Carratala J; SAFO study group. Cloxacillin plus fosfomycin versus cloxacillin alone for methicillin-susceptible Staphylococcus aureus bacteremia: a randomized trial. Nat Med. 2023 Oct;29(10):2518-2525. doi: 10.1038/s41591-023-02569-0. Epub 2023 Oct 2. PMID 37783969
- [Derived] Grillo S, Cuervo G, Carratala J, San-Juan R, Aguado JM, Morata L, Gomez-Zorrilla S, Lopez-Contreras J, Gasch O, Gomila-Grange A, Iftimie S, Garcia-Pardo G, Calbo E, Boix-Palop L, Oriol I, Jover-Saenz A, Lopez-Cortes LE, Euba G, Aguirregabiria M, Garcia-Pais MJ, Gioia F, Pano JR, Pedro-Botet ML, Benitez RM, Perez-Rodriguez MT, Meije Y, Loeches-Yague MB, Horna G, Berbel D, Dominguez MA, Padulles A, Cobo S, Hereu P, Videla S, Tebe C, Pallares N, Miro JM, Pujol M; SAFO study group and the Spanish Network for Research in Infectious Diseases (REIPI). Multicentre, randomised, open-label, phase IV-III study to evaluate the efficacy of cloxacillin plus fosfomycin versus cloxacillin alone in adult patients with methicillin-susceptible Staphylococcus aureus bacteraemia: study protocol for the SAFO trial. BMJ Open. 2021 Aug 5;11(8):e051208. doi: 10.1136/bmjopen-2021-051208. PMID 34353808